CLINICAL TRIAL: NCT04822220
Title: The Effect of Self-Management Program Based on the Individual and Family Self-management Theory on Fatigue, Daily Life Activities and Wellness on Cancer Patients
Brief Title: The Effect of Self-Management Program Based on the Individual and Family Self-management Theory on Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Zeynep KARAKUŞ, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0002
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Oncology; Fatigue; Patient
Keywords: nursing; cancer patients; self-management; fatigue; activities of daily living; well-being; randomized controlled trial
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial consisting of two groups: experimental and control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Fatigue Self-management Programme
  Interventions: Other: Fatigue Self-management Programme
- Controlled (No Intervention): The control group received routine treatment and nursing care

INTERVENTIONS:
Other: Fatigue Self-management Programme — Fatigue Self-management Programme
  Arms: Experimental

SUMMARY:
The purpose of this study is to evaluate the effect of Self-Management Program based on the Individual and Family Self-management Theory on fatigue, daily living activities and well-being of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients for symptom management or supportive care in oncology wards
* Patients who were at first two days of hospitalization
* Patients who had score of 3≤ or ≤7 in Fatigue Visual Analogue Scale (VAS)
* Patients who had score of ≤5 in Pain Analog Visual Scale (VAS)
* Patients who had score of ≤5 The Modified Borg Scale
* Patients who had score of 0, 1, 2 or 3 in ECOG Performance scale
* Patients who had metastases
* Patients who were over 18 years of age
* Patients who had orientation of person, place and time
* Patients who had no communication barriers
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who had hospitalized for the purpose of receiving chemotherapy
* Patients whose Hb value was ≤8 g / dl
* Patients whose body temperature ≥ 38.5 ° C within the last 24 hours
* Patients who had diarrhea in the last 24 hours (frequency of defecation ≥ 3 / day)
* Patients who had a score of ≤ 16 kg / m2 in Body Mass Index (BMI)
* Patients who had advanced heart failure
* Patients who had untreated hypothyroidism
* Patients who diagnosed with major depression and / or treated for depression
* Patients who had no family member involved in their care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in fatigue on the Brief Fatigue Inventory at week 8 | Baseline, 2 week, 4 week, 8 week
  The Brief Fatigue Inventory is a validated, self reported instrument assessing average fatigue.

SECONDARY OUTCOMES:
Change From Baseline in daily living activities on the Katz Index of Independence at week 8 | Baseline, 2 week, 4 week, 8 week
  The Katz Index of Independence is a validated, self reported instrument assessing average daily living activities.
Change From Baseline in well-being on Well-Being Questionnaire (22 items) (W-BQ22) at week 8 | Baseline, 2 week, 4 week, 8 week
  Well-Being Questionnaire (22 items) (W-BQ22) is a validated, self reported instrument assessing average well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Özer, Study Director — Akdeniz University
Locations (1):
- Zeynep Karakuş, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Karakus Z, Ozer Z. The effect of a fatigue self-management program based on individual and family self-management theory in cancer patients: A single-blinded randomized controlled trial. Eur J Oncol Nurs. 2024 Apr;69:102483. doi: 10.1016/j.ejon.2023.102483. Epub 2023 Dec 11. PMID 38417400